CLINICAL TRIAL: NCT05028725
Title: Investigation of a Novel Strategy for Early Detection of Esophageal Squamous Cell Carcinoma
Brief Title: Novel Strategy for Early Detection of Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Johns Hopkins University (Other); Muhimbili University of Health and Allied Sciences (Other); CapNostics, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21457; 5UH3CA211457-04 (NIH); NCI-2021-08885 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Squamous Cell Carcinoma; Esophageal Squamous Dysplasia
Keywords: EsophaCap; Biomarker Detection; Cancer Detection; Chromoendoscopic screening
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Esophageal Squamous Cell Carcinoma (ESCC) Cases (Experimental): Each study participant will undergo esophageal sponge sampling using the 'EsophaCap' sponge device. Group 1 will include a safety-phase, which will consist of a lead-in cohort of 8 patients with ESCC. Subsequent recruitment of ESCC Cases (Group 1) will not commence until the Data Safety Monitoring Board (DSMB) has deemed the safety lead-in data appropriate for continuation. Following collection of esophageal cells, samples will be assessed using the EsoCAN assay. Study participant evaluations will be taken at baseline, immediately after undergoing esophageal sponge sampling, and 7 days following administration of the 'EsophaCap' device.
  Interventions: Device: EsophaCap Sponge; Device: EsoCAN assay
- Non-ESCC, Esophageal squamous dysplasia (ESD) Cases (Experimental): Each study participant will undergo (1) Esophagogastroduodenoscopy (EGD) with chromoendoscopic screening and possible biopsy, and (2) esophageal sponge sampling using the 'EsophaCap' sponge device. Pathology from chromoendoscopic screening will be used to categorize non-ESCC study participants as esophageal squamous dysplasia (ESD) cases and controls. Following collection of esophageal cells, samples will be assessed using the EsoCAN assay. Study participant evaluations will be taken at baseline, immediately after undergoing esophageal sponge sampling, and 7 days following administration of the 'EsophaCap' device.
  Interventions: Device: EsophaCap Sponge; Procedure: Chromoendoscopy; Device: EsoCAN assay
- Non-ESCC, Control Group (Experimental): Each study participant will undergo (1) Esophagogastroduodenoscopy (EGD) with chromoendoscopic screening and possible biopsy, and (2) esophageal sponge sampling using the 'EsophaCap' sponge device. Pathology from chromoendoscopic screening will be used to categorize non-ESCC study participants as esophageal squamous dysplasia (ESD) cases and controls. Following collection of esophageal cells, samples will be assessed using the EsoCAN assay. Study participant evaluations will be taken at baseline, immediately after undergoing esophageal sponge sampling, and 7 days following administration of the 'EsophaCap' device.
  Interventions: Device: EsophaCap Sponge; Procedure: Chromoendoscopy; Device: EsoCAN assay

INTERVENTIONS:
Device: EsophaCap Sponge — Non-invasive strategy to sample esophageal tissue
  Other Names: EsophaCap Sponge Device; EsophaCap Swallowable Sponge device
Procedure: Chromoendoscopy — Lugol's iodine chromoendoscopy is a technique that is used to identify mucosal abnormalities of the esophagus
  Other Names: Lugol's iodine chromoendoscopy; Chromoendoscopic screening
  Arms: Non-ESCC, Control Group; Non-ESCC, Esophageal squamous dysplasia (ESD) Cases
Device: EsoCAN assay — Biomarker Test

SUMMARY:
In the current protocol, we propose a study to evaluate a novel, combined esophageal sponge-methylation biomarker strategy for the early detection of esophageal squamous cell carcinoma (ESCC) as well as its precursor, esophageal squamous dysplasia (ESD). This strategy leverages the 'EsophaCap', a swallowable, retrievable sponge, with subsequent evaluation of the sample using a novel molecular biomarker assay. This biomarker assay evaluates methylation levels in select genes, which have been shown to differ significantly between ESCC cases and controls in pilot studies. Detection of methylation markers highly associated with ESCC could help identify patients with concurrent ESCC or at high risk of imminently developing this condition. If successful, this strategy could result in a paradigm shift for esophageal cancer control strategies in Tanzania and other high-incidence ESCC regions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the sensitivity and specificity of a diagnostic strategy combining esophageal sponge sampling with the 'EsophaCap' sponge device with use of the EsoCAN assay, a novel molecular biomarker assay, among patients with histologically-confirmed ESCC cases and controls.

SECONDARY OBJECTIVES:

I. To evaluate the sensitivity and specificity of a diagnostic strategy combining esophageal sponge sampling with the 'EsophaCap' sponge device with use of the the EsoCAN assay, among patients with histologically-confirmed ESD and controls.

II. To evaluate the safety and feasibility of 'EsophaCap' a swallowable and retrievable sponge, as a non-invasive strategy for screening and early detection of ESCC and its precursor, ESD, in Tanzania.

EXPLORATORY OBJECTIVES:

I. Sensitivity and specificity of esophageal sponge sampling with standard cytological examination among histologically-confirmed ESCC cases and controls.

II. Sensitivity and specificity of esophageal sponge sampling with standard cytological examination among histologically-confirmed ESD cases and controls.

III. To examine methylation levels in new and previously identified genes among patients recruited as suspected ESCC cases who are found to have an alternative diagnosis, with the goal of optimizing the EsoCAN Assay.

OUTLINE:

Each participant will undergo esophageal sponge sampling suing the 'EsophaCap' sponge device. Participants will be on study for up to 38 days.

ELIGIBILITY:
Inclusion Criteria:

ESCC Cases (Group 1):

* Male or female >= 18 years of age at screening visit.
* Patients are currently seen for clinical care at Muhimbili National Hospital (MNH)-Upanga or at MNH-Mloganzila.
* Patient meets one of the following two criteria-
* Patients with a confirmed diagnosis of ESCC as evidenced by histological confirmation OR
* Patient planned to undergo EGD with biopsy for suspected ESCC based upon any one of the following clinical criteria: (1) findings on computed tomography (CT) scan; (2) findings on barium swallow; (3) findings on endoscopy without biopsy confirmation, (4) symptoms of dysphagia and/or odynophagia without an alternative explanation for these symptoms.
* Patient must be able to swallow liquid (Ogilvie's score < 3).
* Patients must be well enough to participate in a 20-minute interview or have a close relative who is able to do so on their behalf.
* Patients must be willing to be contacted either in person or via phone 7-10 days following administration of the 'EsophaCap' sponge device.
* Native of Tanzania.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Non-ESCC study participants (Group 2):

* Male or female ≥ 18 years of age at screening visit.
* Patients are currently seen for clinical care at MNH-Upanga or at MNH-Mloganzila.
* Patient is scheduled to undergo EGD for a suspected non-malignant condition with no symptoms concerning for esophageal cancer (i.e. dysphagia or odynophagia).
* Patient must be able to swallow liquid (Ogilvie's score < 3).
* Patients must be well enough to participate in a 20-minute interview or have a close relative who is able to do so on their behalf.
* Patients must be willing to be contacted either in person or via phone 7-10 days following administration of the 'EsophaCap' sponge device.
* Native of Tanzania.
* Written informed consent (and assent when applicable) obtained from participant or participant's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

ESCC Cases (Group 1):

* Known pregnancy during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Clinical instability (i.e. hypotension or a recent cardiovascular event).
* Any history of upper gastrointestinal bleeding within the past 3 months (including reported history of hematemesis and/or melena).
* Diagnosis of peptic ulcer disease within the last 3 months.
* Known history of esophageal varices.
* Patients taking anticoagulation or antiplatelet therapy/medication (warfarin, clopidogrel, aspirin, heparin or enoxaparin) for high-risk conditions.
* Patients with an active extra-esophageal malignancy (not currently in remission).
* Patient with a known history of a non-malignant esophageal stricture.
* Patients with esophageal stents currently in place.
* Patients with a history of radiation therapy to the head, neck, any part of the gastrointestinal tract (including esophagus) or thorax.
* Patients who have previously received chemotherapy in the last 12 months
* Patients with any history of major surgery for esophageal cancer (e.g. esophageal bypass, esophagectomy, etc.).
* Patients who have a known history of or clinical symptoms concerning for tracheoesophageal fistula (aspiration history, severe cough)
* Patients with a known history of small bowel obstruction
* Patients with a history of bleeding complications during esophageal biopsy.
* Patients with any history of a head and neck malignancy.
* Patients with a known bleeding disorder
* Patients with known thrombocytopenia (less than 50,000 platelets per microliter)
* Individuals who are not permanent residents or natives of Tanzania.
* Inability to follow instructions.
* Unable to provide informed consent.

Non-ESCC study participants (Group 2):

* Known pregnancy during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Clinical instability (i.e. hypotension or a recent cardiovascular event).
* Any history of upper gastrointestinal bleeding within the past 3 months (including reported history of hematemesis and/or melena).
* Diagnosis of peptic ulcer disease within the last 3 months.
* Known history of esophageal varices.
* Patients taking anticoagulation or antiplatelet therapy/medication (warfarin, clopidogrel, aspirin, heparin or enoxaparin) for high-risk conditions.
* Patients with an active extra-esophageal malignancy (not currently in remission) or any history of a non-cutaneous malignancy diagnosed within the previous five years.
* Patient with a known history of esophageal strictures disabling passage of the capsule.
* Patient with esophageal stents currently in place.
* Patients with a history of radiation therapy to the head, neck, any part of the gastrointestinal tract (including esophagus) or thorax.
* Patients with a known history of small bowel obstruction
* Patients with a known bleeding disorder
* Patients with known thrombocytopenia (less than 50,000 platelets per microliter)
* Individuals who are not permanent residents or natives of Tanzania.
* Allergy to iodine
* Presence of goiter.
* Inability to follow instructions.
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of True-Positives (sensitivity) detected with the EsoCAN assay after specimen collection using 'EsophaCap' sponge sampling (ESCC cases & controls only) | Up to 38 days
  The proportion of participants with a positive EsoCAN assay result, among patients with histologically-confirmed Esophageal Squamous Cell Carcinoma (ESCC). The following equation will be used as a cut point for ESCC using the EsoCAN assay [0.139*log2(gene A)] + [0.176* log2(gene B)] + [0.185* log2(gene C)], whereas a cutoff value (for the numerical index produced by this formula) of greater than -2.327 is classified as positive.
Proportion of True-Negatives (specificity) detected with the EsoCAN assay after specimen collection using 'EsophaCap' sponge sampling (ESCC cases & controls only) | Up to 38 days
  The proportion of participants with a negative EsoCAN assay result for will be reported, among study participants who are classified as controls. The following equation will be used as a cut point for ESCC using the EsoCAN assay [0.139*log2(gene A)] + [0.176* log2(gene B)] + [0.185* log2(gene C)], whereas a cutoff value (for the numerical index produced by this formula) of less than -2.327 is classified as negative.

SECONDARY OUTCOMES:
Proportion of True-Positives (sensitivity) detected with the EsoCAN assay after specimen collection using 'EsophaCap' sponge sampling (ESD cases & controls only) | Up to 38 days
  The proportion of participants with both a positive EsoCAN assay result, among patients with histologically-confirmed Esophageal Squamous Dysplasia (ESD). The following equation will be used as a cut point for ESD: [0.139*log2(gene A)] + [0.176* log2(gene B)] + [0.185* log2(gene C)], whereas a cutoff value (for the numerical index produced by this formula) of greater than -2.327 is classified as positive.
Proportion of True-Negatives (specificity) detected with the EsoCAN assay after specimen collection using 'EsophaCap' sponge sampling (ESD cases & controls only) | Up to 38 days
  The proportion of participants with a negative EsoCAN assay result will be reported. The following equation will be used as a cut point for ESD: [0.139*log2(gene A)] + [0.176* log2(gene B)] + [0.185* log2(gene C)], whereas a cutoff value (for the numerical index produced by this formula) of less than -2.327 is classified as negative.
Proportion of study participants who successfully swallow the esophageal sponge device | Up to 38 days
  The success of swallowing the esophageal sponge device will be determined by the clinical team overseeing the EsophaCap' administration and categorized as a dichotomous response of Yes (successful) or No (not successful).
Proportion of study participants who experienced an esophageal sponge device-related adverse event in the lead in cohort of ESCC Cases | Up to 38 days
  Adverse events for the lead in cohort with histologically confirmed or suspected ESCC based upon pre-specified clinical criteria will be reported and graded and classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Median Acceptability Scores | Up to 38 days
  Participants will be asked to rate their satisfaction with their experience with the EsophaCap sponge procedure after the procedure is complete by selecting a score on a scale with corresponding facial images with scores ranging between 0='Best Experience' (large smile on facial expression) to 10='Worst experience' (crying and frowning facial expression).

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Buckle, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- Tanzania (2):
  - Muhimbili National Hospital (MNH), Dar es Salaam, Mloganzila
  - Muhimbili National Hospital (MNH), Dar es Salaam, Upganda

IPD SHARING:
Plan to Share IPD: No